CLINICAL TRIAL: NCT03950661
Title: Walking Green: The Effects of Walking in Forested and Urban Areas on Health and Well-being
Brief Title: Walking Green: The Effects of Walking in Forested and Urban Areas
Acronym: NUWG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00201604
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Mood; Stress; Anxiety; Depression; Obesity; Health Behavior; Physical Activity
Keywords: nature; walk; stress; Green Walking; Physical Activity; Environment; anxiety; mood
MeSH Terms: conditions — Anxiety Disorders; Depression; Obesity; Health Behavior; Motor Activity | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Randomized cross over design. Repeated measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forest (Experimental): Each subject is exposed to a 50 minute walk in a "green location" at some point during the crossover experiment. The psychological and physiological measurements taken during these walk location weeks are compared to the measurements from the other location. In addition a 'control' day is assigned for each location (ADL).
  Interventions: Other: Walking
- Urban (Experimental): Each subject is exposed to a 50 minute walk in a "gray location" at some point during the crossover experiment. The psychological and physiological measurements taken during these walk location weeks are compared to the measurements from the other location. In addition a 'control' day is assigned for each location (ADL).
  Interventions: Other: Walking

INTERVENTIONS:
Other: Walking

SUMMARY:
This research hypothesizes that moderate physical activity in a "green environment" (e.g. a forest preserve path) has increased benefits on psychological measures (stress, anxiety, mood, depression, attention) and on physiological measures (Heart Rate Variability, Blood Glucose, Salivary Cortisol) when directly compared to activity in a "gray environment" (urban or suburban sidewalks).

The study design is a randomized crossover design in which each subject is assigned randomly to a group which determines the order in which participants will walk in each location. Subjects will take three 50-minute walks per location in one week, with half of the subjects taking the urban walks first as per group assignment. Control data are collected on days when participants do not walk. Physiological data are taken during walks and control periods (heart rate, heart rate variation). Biomarker samples (saliva, dried blood spots) are taken on selected days. Psychological data are take before and after walks and control periods.

DETAILED DESCRIPTION:
This study records the psychological and physiological effects of green vs gray walks during a longitudinal crossover study on 41 participants. In accordance with the Attention Restoration and Stress Recovery theories we hypothesize that exposure to a green environment will have beneficial health outcomes for participants both psychologically (mood, stress, anxiety, depression, attention) and physiologically (blood glucose, heart rate variability, cortisol).

Participants will be randomly assigned to a study group which determines the order in which they will walk in either the gray or green location. The study takes place for 29 days of which only 9 are active study dates. The cross-over design controls for training effects that may result from the regular physical activity. Participants provided informed consent on Day 1. Walks will be monitored on Days 8, 12, 22, 26, while walks on days 10 and 24 have no monitoring to reduce testing burden. Days 15 and 29 are control days in which the participants are monitored during the day (Activities of Daily Living) as a control against the location they had previously walked in. No walks will be taken between days 12 and 21 to provide a washout period from the previous location. Psychological tests are administered by computer using the Qualtrics software platform to assess:

Positive and Negative Affect Scale (PANAS) Center for Epidemiological Studies Depression Scale (CESD) State and Trait Anxiety Inventory (STAI) Cohen's Perceived Stress Scale (UCLA) Perceived Isolation Scale Nature Relatedness Scale (NR-6)

Anthropometric measures are taken on days 1, 8, 15, 22, and 29. Physiological effects are studied through heart rate monitoring during all monitored walks via a Zephyr Omnisense which records heart information as well as activity, temperature and breathing rate. Salivary cortisol is collected on days 7, 14, 21, and 28 by the participant. Blood glucose is measured on days 8, 12, 15, 22, 26, and 29; dried blood spots are collected for future analysis of inflammatory biomarkers.

Hypotheses will be tested using fixed and random effects linear regression models using the appropriate statistical procedures in SAS 9.4 to test for main effects, covariates, and other confounding variables that were measured throughout the study including individuals' reported stress and tiredness, and the weather conditions of the day.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* under the age of 35
* no current infections / recent infections (<2weeks)
* PAR-Q+ scores indicative of readiness to engage in physical activity

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Inability to consent
* Incarcerated Persons
* non-adults

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Psychological Effects - Mood | 29 days
  Change in Positive and Negative Affect scale 0 = never, 4 = very often. Higher Positive Affect scores reflect better reported mood scores. Lower Negative Affect Scores reflect better mood scores. Average values based on age
Psychological Effects - Anxiety | 29 days
  change in STAI (STAI-TRAIT anxiety) score based on a Likert scale self reported score. Higher scores indicate a higher level of self-reported anxiety.
Psychological Effects - Attention | 29 days
  change in vBDS (backward digit span) score lower scores indicate a increased inability to properly recall the numbers in the test.
Psychological Effects - Depression | 29 days
  change in CESD score. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology. Citation: Radloff LS: The CES-D Scale: a self-report depression scale for research in the general population.

SECONDARY OUTCOMES:
Physiological Effects - Blood Glucose | 29 days
  Glucose levels as markers of health and wellness. (mg/dL)
Physiological Effects - Salivary Cortisol | 29 days
  Diurnal cortisol dynamics measured by salivary cortisol (ug/dl), as the normal drop in cortisol during the day is attenuated by exposure to chronic stress.
Physiological Effects - Blood | 29 days
  Pro- and anti-inflammatory cytokine concentrations in blood (pg/mL), as stress typically induces an inflammatory response
Physiological Effects - Heart Rate Variation | 29 days
  changes in HRV is indicative of parasympathetic input (milliseconds), higher HRV correlating to reduced stress.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Horton, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No